CLINICAL TRIAL: NCT06732570
Title: Effect of High Intensity Laser on Shoulder Impingement Syndrome in Adolescents
Brief Title: Effect of High Intensity Laser on Shoulder Impingement.
Acronym: lasershoulder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd Elkhalek Mansour Ahmed, physical therapist, Al Azhar university hospital, MSC, DPT, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: high power laser for shoulder
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: High Intensity Laser; Shoulder Impingement Syndrome; Shoulder Pain
Keywords: high intensity laser, shoulder impingement, manual therapy, exercise therapy, shoulder dysfunction; shoulder function; pain; adolescents
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Pain | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Pretest posttest randomized controlled trail.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- group A: manual therapy and exercise (Active Comparator): will receive the therapeutic exercises (rotator cuff strengthening, cools ex's, serratus punch ex, pectoralis minor flexibility and posterior capsule modified sleeper stretching ex's) and manual therapy (mulligan abduction, deep transverse friction technique on the supraspinatus muscle, scapular mobilization, caudal and posterior humeral mobilization), they will receive 15 consecutive sessions (three session weekly over 5 weeks).
  Interventions: Other: manual therapy; Other: exercise therapy
- group (B): high intensity laser, manual therapy, exercise therapy (Experimental): will receive high intensity laser therapy (PAGANI scanner 16 j/cm2, high power laser BI-POWER SN/ 477 made in Italy will be used)three sessions weekly over 5 weeks. the patient will be in supine position with shoulder uncovered from clothes and wearing laser protective eye glass, the dose will be selected from device pathologies list programs number thirty-four with 30% power, frequency continuous, density 16 j/cm2, time automatically adjusted by the device according to the width of scanning area ( superiorly from the acromioclavicular joint down to end of biceps tendon and medially from the coracoid process to the middle fiber of deltoid laterally) and the infrared will be ON.
  therapeutic exercises (rotator cuff strengthening, cools ex's, serratus punch ex, pectoralis minor flexibility and posterior capsule modified sleeper stretching ex's) and manual therapy (mulligan abduction, deep transverse friction on supraspinatus, scapular mobilization, caudal and posterior humerla glide)
  Interventions: Device: high intensity laser; Other: manual therapy; Other: exercise therapy

INTERVENTIONS:
Device: high intensity laser — the patient will be in supine position with shoulder uncovered from clothes and wearing laser protective eye glass to protect eye from laser radiation, the dose will be selected from device pathologies list programs number thirty-four with 30% power, frequency continuous, density 16 j/cm2, time automatically adjusted by the device according to the width of scanning area ( superiorly from the acromioclavicular joint down to end of biceps tendon and medially from the coracoid process to the middle fiber of deltoid laterally) and the infrared will be ON.
  Arms: group (B): high intensity laser, manual therapy, exercise therapy
Other: manual therapy — manual therapy (mulligan shoulder abduction, deep transverse friction technique on the supraspinatus tendon, scapular mobilization, caudal and posterior humeral mobilization) three session weekly over 5 weeks.
Other: exercise therapy — therapeutic exercises (rotator cuff strengthening, cools ex's, serratus punch supine ex, pectoralis minor flexibility (focused and gross stretch) and posterior capsule modified sleeper stretching ex's from side)

SUMMARY:
Treatment for shoulder impingement is conservative initially, Rehabilitation programs generally consist of exercise therapy and manual therapy that provide relief from symptoms of impingement. High-intensity laser therapy used recently and was found to be effective in the short term in the treatment of pain and disability in patients with impingement.

This study aims to

* Investigate the effect of high intensity power laser therapy on sonographic measurement in the adolescent suffering from shoulder impingement syndrome.
* Investigate the effect of high intensity power laser therapy on pain in the adolescent suffering from shoulder impingement syndrome.
* Investigate the effect of high intensity power laser therapy on shoulder function in the adolescent suffering from shoulder impingement syndrome.

RESEARCH QUESTION:

Does using high intensity power laser affects shoulder dysfunction in adolescent with shoulder impingement syndrome?

DETAILED DESCRIPTION:
Shoulder symptoms are often persistent and recurrent and represents approximately one fifth of all musculoskeletal disability payment. One of the most common causes of shoulder pain is the occurrence of tendinopathy resulting from the impingement of rotator cuff tendons under the coracoacromial arch which refer to impingement syndrome.

Treatment for shoulder impingement is conservative initially, Rehabilitation programs generally consist of exercise therapy that provide relief from symptoms of impingement, Exercise therapy has been shown to be effective in the reducing pain and improving function also it was stated that the exercise therapy lead to improving shoulder musculoskeletal risk factors in competitive athletes with Specific exercise was superior to non-specific exercise. Strong recommendation may be made to include manual therapy as an adjunct intervention with exercise.

The manual therapy technique of joint mobilizations which are commonly used by physiotherapists for reducing pain and disability in patients with shoulder musculoskeletal disorders, Manual therapy which involves realigning collagen, enhancing fiber slip, reducing adhesion, and re-establishing correct gleno-humeral joint kinematics, can relieve pain by stimulating peripheral mechanical receptors, suppressing nociceptors, boosting synovial fluid nutrition, and reducing adhesion. It has been stated that impingement patients treated with manual therapy in combination with supervised exercise showed improvement in pain and function.

High-intensity laser therapy (HILT) is a treatment method that added to therapeutic interventions recently. HILT improves the microcirculation and tissue regeneration with photomechanic effects in deep tissues. Biostimulation, anti-inflammatory, and analgesic properties contribute to an effective improvement in painful bone-muscle-joint pathologies, including shoulder problems. Adding therapeutic interventions to laser therapy is usual in clinical practice. HILT was found to be effective in the short term in the treatment of pain and disability in patients with Sub-acromial pain syndrome.

Ultrasonography is recommended as the first line imaging tool to evaluate sports injuries; it has been used as the preferred technique for evaluating the subacromial space.

Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. . This technique is a well-known and well-validated method to induce acute experimental pain.

Null Hypothesis:

High intensity laser therapy will not affect the sonographic measurement in adolescents with shoulder impingement syndrome.

High intensity laser therapy will not affect the pain in adolescents with shoulder impingement syndrome.

High intensity power laser therapy will not affect the shoulder function in adolescents suffering from shoulder impingement syndrome.

Basic assumptions:

It will be assumed that:

* All evaluation and treatment procedures will be performed in the same environment for all patients
* All volunteers will attend the treatment program regularly.
* All volunteers will be cooperative, following the instructions given to them, and exert their maximum effort during the study.
* The results of the study will be helpful for physical therapists dealing with similar cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age was ranged between 12-18 years old.
2. Unilateral pain in the anterolateral region of the shoulder.
3. Has painful arc.
4. 2 out of 3 impingement tests positive (Hawkins, Jobe and Neer).
5. Pain with palpation of the supraspinatus tendon insertion.

Exclusion Criteria:

1. Previous shoulder complex, cervical and thoracic fractures, or surgeries.
2. Either cervical pain or arm radiculopathy.
3. History of shoulder dislocation.
4. Traumatic onset of the pain.
5. No corticosteroid injections could have been received within 2 months prior to the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acromio-humeral distance (AHD) and Coraco-humeral distance (CHD). | measurements will be done pre and post 5 weeks (15 sessions, three sessions per week) of interventions.
  Musculoskeletal Ultrasound (TOSHIBA Aplio 500, japan. Linear probe 12-15 MHZ) will be used to measure both distance (AHD& CHD) with the injured shoulder in two angles 0- and 60-degrees abduction from scapular plane (40° front of the frontal plane). The subjects were instructed to sit upright in the chair and to place their feet on the floor with knees and hips 90 degrees flexion. the examiner took one ultrasound image at angle 0-degree abduction as thepatient's arm rest beside the body with the palm toward the body and the other image from 60 abduction from scaption. acromio-humeral distance calculated by measuring the linear distance from the most lateral edge of the acromion to the most proximal portion of the humeral head. Then for calculation of the coraco-humeral distance the ultrasound transducer was placed over the most anterior aspect of the shoulder, observing the coracoid process and the humeral head on the screen, taking the shortest distance between them (in centimeters).
pain. | measurements will be done pre and post 5 weeks (15 sessions, three sessions per week) of interventions.
  pain: BASLINE push pull force gauge algometer (White Plains, New York 10602 USA) will be used to assess patient pain. An algometer can be used to objectively measure the first point of pressure required to produce symptoms at the most painful points in the long head of biceps tendon, under acromion area and deltoid with the patient relaxed and the affected shoulder will be uncovered from clothes.
Function. | measurements will be done pre and post 5 weeks (15 sessions, three sessions per week) of interventions.
  Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability which take less than five minutes to complete. The examiner will describe to the patient the two scale parts, the pain scale that is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage. A score of 0 indicates best, 100 indicates worst. A higher score shows more disability. In scoring SPADI, any question missed should be taken out of the total score of each subscale. i.e if 1 question is omitted in the pain section, the total score is divided by 40.

CONTACTS AND LOCATIONS:
Overall Officials: Abd ELkhalek Mansour Ahmed, MSC, DPT, Study Director — physical therapist, Al Azhar university hospital, Sayed Galal hospital; Khaled Ahmed olama, professor, Study Director — Physical Therapy, Department for Physical Therapy for pediatrics Faculty of Physical Therapy Cairo University; mohamed Ali Elshafey, professor, Study Director — Physical Therapy, Department for Physical Therapy for pediatrics Faculty of Physical Therapy Cairo University; hatem Mohamed El-Azizi, professor, Study Director — Radiology Department, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided